CLINICAL TRIAL: NCT03563027
Title: Evaluating Connected Health Approaches to Improving the Health of Veterans (CDA 15-065)
Brief Title: Social and Financial Incentives to Increase Physical Activity Among Overweight and Obese Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CDX 18-003; HX-001922-01 (Other Grant/Funding Number: Cpl Michael J. Crescenz VA Medical Center)
Record Dates: First submitted 2018-06-06; First posted 2018-06-20 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Physical Activity
Keywords: Physical activity; Incentive; Wearable device; Gamification
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel 3-arm randomized, controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes assessor will be masked until the trial is completed and all analyses are finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): This arm serves as control and uses a wearable device to track daily step counts
- Social Incentive Gamification (Experimental): This arm uses a wearable device to track daily step counts, is entered into social incentive gamification, and selects a support sponsor
  Interventions: Behavioral: Social Incentive Gamification; Behavioral: Support Sponsor
- Social Incentive Gamification and Financial Incentive (Experimental): This arm uses a wearable device to track daily step counts, is entered into social incentive gamification, selects a support sponsor, and receives a financial incentive
  Interventions: Behavioral: Social Incentive Gamification; Behavioral: Support Sponsor; Behavioral: Financial Incentive

INTERVENTIONS:
Behavioral: Social Incentive Gamification — Game-based intervention with points and levels
  Arms: Social Incentive Gamification; Social Incentive Gamification and Financial Incentive
Behavioral: Support Sponsor — Participants select a support sponsor to receive weekly updates on progress in the game
  Arms: Social Incentive Gamification; Social Incentive Gamification and Financial Incentive
Behavioral: Financial Incentive — Participants receive a loss-framed financial incentive allocated upfront each week and financial incentives taken away each day the goal is not met
  Arms: Social Incentive Gamification and Financial Incentive

SUMMARY:
In this randomized, controlled trial the investigators will compare the use of social and financial incentive-based interventions to increase physical activity among overweight and obese Veterans during a 12-week intervention with 8 weeks of follow-up.

DETAILED DESCRIPTION:
In this 3-arm randomized trial, the investigators will compare the effectiveness of a social incentive-based gamification intervention with and without loss-framed financial incentives to increase physical activity relative to a control among overweight and obese adults Veterans. All Veterans will use a Fitbit wearable device to establish a baseline step count, select a step goal increase of 33% to 50% above baseline and then participate in a 12-week intervention and 8-week follow-up period. The two intervention arms will be entered into a game with points and levels designed using insights from behavioral economics. They will be asked to select a social support partner who will receive weekly updates on their progress in the game. Veterans in one arm will also receive loss-framed financial incentives allocated to an account each week during the intervention and financial incentives taken away each day the step goal was not achieved.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Body mass index of 25 or greater
* Access to smartphone or tablet to sync wearable device data
* Interest in participating in a 20-week physical activity program

Exclusion Criteria:

* Already participating in a physical activity research study
* Unable to provide informed consent
* Unsafe or infeasible to participate
* No access to smartphone or table to sync wearable device data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S. Patel, MD MBA MS, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal AK, Waddell KJ, Small DS, Evans C, Harrington TO, Djaraher R, Oon AL, Patel MS. Effect of Gamification With and Without Financial Incentives to Increase Physical Activity Among Veterans Classified as Having Obesity or Overweight: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116256. doi: 10.1001/jamanetworkopen.2021.16256. PMID 34241628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
Started | 60 | 60 | 60
Completed | 60 | 60 | 58
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 44 | 39 | 122
  >=65 years | 21 | 16 | 21 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.6) | 53.7 (13.0) | 57.9 (12.6) | 56.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 20 | 71
  Male | 38 | 31 | 40 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 5 | 13
  Not Hispanic or Latino | 55 | 52 | 52 | 159
  Unknown or Not Reported | 0 | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 60 | 180
Weight, lbs. [Mean (Standard Deviation); unit: Pounds] | 216.7 (41.9) | 218.1 (47.8) | 217.1 (35.2) | 217.3 (41.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 32.6 (5.1) | 33.7 (6.3) | 32.8 (5.4) | 33.0 (5.6)
Baseline Step Count [Mean (Standard Deviation); unit: Daily step count] | 5881 (2038) | 6012 (2494) | 6105 (2320) | 6000 (2300)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Steps From Baseline Relative to Control
Description: Daily steps counts
Time Frame: Intervention period of weeks 5 to 12 which excludes the 4-week ramp-up
Measure: Mean (Standard Deviation); unit: Mean daily steps
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
Number analyzed (Participants) | 60 | 60 | 58
Mean daily steps | 6195 (3767) | 6709 (3827) | 7599 (3897)
Statistical Analysis 1: Comparison: Control vs Social Incentive Gamification; Test type: Superiority; p = .81, Regression, Linear; Mean Difference (Net) = 433, 95% CI 2-sided [-337 to 1203]
Statistical Analysis 2: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p = .005, Regression, Linear; Mean Difference (Net) = 1224, 95% CI 2-sided [451 to 1996]

2. Secondary Outcome: Change in Mean Daily Steps From Baseline Relative to Control
Description: Daily step counts
Time Frame: Follow-up period of weeks 13 to 20
Measure: Mean (Standard Deviation); unit: Mean daily steps
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
Number analyzed (Participants) | 60 | 60 | 58
Mean daily steps | 6272 (3839) | 6213 (3666) | 6962 (3888)
Statistical Analysis 1: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p = .92, Regression, Linear; Mean Difference (Net) = -160, 95% CI 2-sided [-983 to 663]
Statistical Analysis 2: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p = .37, Regression, Linear; Mean Difference (Net) = 564, 95% CI 2-sided [-261 to 1389]

3. Secondary Outcome: Proportion of Participant-days Step Counts Were Achieved Relative to Control
Description: Proportion of days for a participants that their step goal target was achieved
Time Frame: Intervention period of weeks 5 to 12 which excludes the 4-week ramp-up
Measure: Mean (Full Range); unit: Proportion of participant days
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
Number analyzed (Participants) | 60 | 60 | 58
Proportion of participant days | .25 [0 to 1.0] | .41 [0 to 1.0] | .48 [0 to 1.0]
Statistical Analysis 1: Comparison: Control vs Social Incentive Gamification; Test type: Superiority; p < .001, Regression, Linear; Median Difference (Net) = .21, 95% CI 2-sided [.18 to .24]
Statistical Analysis 2: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p < .001, Regression, Linear; Mean Difference (Net) = .34, 95% CI 2-sided [.31 to .37]

4. Secondary Outcome: Proportion of Participant-days Step Counts Were Achieved
Description: Proportion of days for a participants that their step goal target was achieved
Time Frame: Follow-up period of weeks 13 to 20
Measure: Mean (Full Range); unit: Proportion of participant days
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
Number analyzed (Participants) | 60 | 60 | 58
Proportion of participant days | .26 [0 to 1.0] | .32 [0 to 1.0] | .37 [0 to 1.0]
Statistical Analysis 1: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p < .001, Regression, Linear; Mean Difference (Net) = .09, 95% CI 2-sided [.06 to 0.1]
Statistical Analysis 2: Comparison: Control vs Social Incentive Gamification and Financial Incentive; Test type: Superiority; p < .001, Regression, Linear; Median Difference (Net) = .18, 95% CI 2-sided [.15 to .20]

ADVERSE EVENTS:
Time Frame: 22 weeks
Arm/Group | Control | Social Incentive Gamification | Social Incentive Gamification and Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
First, participants were from a single VA system and needed access to a smartphone or tablet, which may limit generalizability. Second, among the 10,000 Veterans invited by mail, only about 7% expressed interest and only about 2% were ultimately enrolled. These participants had higher than step counts at baseline and may not be representative of the target population for this type of intervention. Third, we evaluated activity using step counts, did not have data on other measures of activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT03563027/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03563027/SAP_001.pdf